CLINICAL TRIAL: NCT06177925
Title: A Phase Ⅱ Exploratory Clinical Study of Adebrelimab Combined With Chemotherapy and Concurrent Radiotherapy as First-Line Treatment for Extensive-Stage Oligometastatic Small Cell Lung Cancer
Brief Title: A Phase Ⅱ Clinical Study of Adebrelimab Combined With Chemotherapy and Concurrent Radiotherapy for Extensive-Stage Oligometastatic SCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2023-465
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Carcinoma, Bronchogenic; Bronchial Neoplasms; Lung Neoplasms; Small Cell Lung Carcinoma
Keywords: Extensive stage small cell lung cancer; Oligometastasis; Adebrelimab; Chemotherapy; Radiotherapy
MeSH Terms: conditions — Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Carcinoma, Bronchogenic; Bronchial Neoplasms; Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Carboplatin; Cisplatin; Etoposide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Adebrelimab, chemotherapy, radiation therapy) (Experimental): Participants will receive Adebrelimab intravenously in combination with carboplatin /Cisplatin and etoposide during the induction phase (2 Cycles ). Thereafter, participants will receive concurrent chemoradiotherapy(thoracic radiation therapy and SBRT for metastases,combination with carboplatin /Cisplatin and etoposide for 1-2 Cycles).Then participants will receive Adebrelimab combination with carboplatin /Cisplatin and etoposide for 1-2 Cycles,followed by Adebrelimab maintenance until persistent radiographic PD, intolerable toxicity or withdrawal of consent during the maintenance phase.
  Interventions: Drug: Adebrelimab; Drug: Carboplatin/Cisplatin; Drug: Etoposide; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Adebrelimab — Adebrelimab intravenous infusion will be administered during the induction phase (Cycles 1-2 ) and maintenance phase.
Drug: Carboplatin/Cisplatin — Carboplatin/Cisplatin intravenous infusion will be administered during the induction phase, concurrent chemoradiotherapy phase and maintenance phase(Cycles 1-4 or 6).
Drug: Etoposide — Etoposide intravenous infusion will be administered during the induction phase, concurrent chemoradiotherapy phase and maintenance phase(Cycles 1-4 or 6).
Radiation: Radiation therapy — IMRT for thoracic of 45--55Gy in 15-22 fractions，SBRT for metastases during the concurrent chemoradiotherapy phase

SUMMARY:
This is an open-label, single arm Phase II study designed to evaluate the efficacy and safety of adebelizumab combined with carboplatin/Cisplatin plus (+) etoposide and concurrent radiotherapy in the first-line treatment of patients with extensive stage oligometastatic small cell lung cancer.

DETAILED DESCRIPTION:
Participants will receive Adebrelimab intravenously in combination with carboplatin /Cisplatin and etoposide during the induction phase (2 Cycles ). Thereafter, participants will receive concurrent chemoradiotherapy(thoracic radiation therapy and SBRT for metastases,combination with carboplatin /Cisplatin and etoposide for 1-2 Cycles).Then participants will receive Adebrelimab combination with carboplatin /Cisplatin and etoposide for 1-2 Cycles,followed by Adebrelimab maintenance until persistent radiographic PD, intolerable toxicity or withdrawal of consent during the maintenance phase.

ELIGIBILITY:
Inclusion Criteria:

* Signed inform consent form
* Age >= 18 years and <= 75 years
* Histologically or cytologically confirmed ES-SCLC (per the Veterans Administration Lung Study Group [VALG] staging system)，the number of metastatic lesions ≤ 5, the number of metastatic organs ≤ 3, and no previous systemic chemotherapy, radiotherapy or immune checkpoint inhibitor treatment.
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Expected survival time ≥ 3 months
* Patients must submit a pre-treatment tumor tissue sample during the study.
* Adequate hematologic and end organ function

Exclusion Criteria:

* Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for ≥ 1 week prior to randomization
* Leptomeningeal disease
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
* Uncontrolled or symptomatic hypercalcemia
* Malignancies other than SCLC within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome
* History of autoimmune disease, including but not limited to myasthenia gravis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease
* Prior treatment with immune checkpoint blockade therapies
* Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of first administration of study treatment. Inhaled or topical steroids, and adrenal replacement steroid are permitted in the absence of active autoimmune disease.
* Significant cardiovascular disease
* Prior allogeneic bone marrow transplantation or solid organ transplant
* Treatment with systemic immunosuppressive medications within 1 weeks prior to randomization
* History of hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins, carboplatin or etoposide
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-12-10 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | up to approximately 30 months

SECONDARY OUTCOMES:
Overall Survival (OS) | up to approximately 30 months
Objective Response Rate (ORR) | up to approximately 30 months
Disease control rate (DCR) | up to approximately 30 months
Duration of Response (DOR) | up to approximately 30 months
Percentage of Participants Alive at 1 Year and 2 Years | 1 year, 2 years
Percentage of Participants Alive and Without PD at 6 Months and 1 Year | 6 months, 1 year
Percentage of Participants with Adverse Events Or Serious Adverse Events | up to approximately 30 months

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No